CLINICAL TRIAL: NCT03843710
Title: A Phase 2, Pilot Open Label, Sequential Group, Investigator Blinded Study of Magnetic Resonance Spectroscopy (31P-MRS) to Assess the Effects of CNM-Au8 for the Bioenergetic Improvement of Impaired Neuronal Redox State in Amyotrophic Lateral Sclerosis
Brief Title: 31P-MRS Imaging to Assess the Effects of CNM-Au8 on Impaired Neuronal Redox State in Amyotrophic Lateral Sclerosis (REPAIR-ALS)
Acronym: REPAIR-ALS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study execution discontinued at this time.
Sponsor: Clene Nanomedicine (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNMAu8.203
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Neurodegeneration; gold; nanocrystal; NAD+; NADH; Redox; Redox Ratio; ALS; Amyotrophic Lateral Sclerosis; 31P-MRS; MRS; magnetic resonance spectroscopy; nanoparticle; nanomedicine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: Open Label, Investigator Blinded, Sequential Cohort (max of 2 cohorts amongst the possible 4 interventions)
Masking Description: Research participants and site personnel are not masked to study drug, but will be blinded to study dose for each cohort (single-blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 7.5mg CNM-Au8 (Experimental): 7.5mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals
- 15mg CNM-Au8 (Experimental): 15mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals
- 30mg CNM-Au8 (Experimental): 30mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals
- 60mg CNM-Au8 (Experimental): 60mg suspension of clean-surfaced, faceted, gold nanocrystals in 120ml of sodium bicarbonate buffered water
  Interventions: Drug: Gold Nanocrystals

INTERVENTIONS:
Drug: Gold Nanocrystals — CNM-Au8 is a dark red/purple-colored liquid formulation consisting of a stable suspension of faceted clean surfaced elemental gold nanocrystals in buffered deionized water with a concentration of up to 0.5 mg/mL of gold. The formulation is buffered by sodium bicarbonate present at a concentration of 0.546 mg/mL. There are no other excipients. The drug product is formulated to be taken orally and will be provided in single dose HDPE containers. The study doses vary by the concentration of gold nanocrystals per milliliter in a volume of 60 mL.
  Other Names: CNM-Au8

SUMMARY:
REPAIR-ALS is a single-center open label pilot, sequential group, investigator and patient blinded study to assess the CNS metabolic effects, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who have been diagnosed with Amyotrophic Lateral Sclerosis (ALS) within twelve (12) months of Screening. The primary endpoint is the ratio of the oxidized to reduced form of nicotinamide adenine dinucleotide (NAD+:NADH) measured non-invasively by 31phosphorous magnetic resonance spectroscopy (31P-MRS).

DETAILED DESCRIPTION:
This is a single-center open label pilot, sequential group, investigator blinded study of the CNS metabolic effects, safety, pharmacokinetics, and pharmacodynamics of CNM-Au8 in patients who have been diagnosed with Amyotrophic Lateral Sclerosis within twelve months of Screening. The Sponsor will select a starting treatment dose of CNM-Au8 for the initial treatment. Investigators and patients will be blinded to each cohort's study dose. Upon completion of the first treatment cohort, the Sponsor will select a single dose or two different doses for the subsequent second cohort from a pre-specified dosing selection plan based on the evaluation of the 31P-Magnetic Resonance Spectroscopy (31P-MRS) changes versus baseline in the first cohort. Up to a total of two treatment cohorts may be studied (n=12 patients/cohort, total n=24 patients). All patients will receive daily oral treatment over twelve consecutive weeks during each cohort's Treatment Period.

There will be three study periods per treatment cohort:

A four-week screening period (Screening Period); A twelve-week treatment period (Treatment Period); A four-week follow-up period (End-of-Study Assessment).

The primary study outcome, CNS metabolic changes, will be assessed based upon each patient's Week 12 study visit versus the pre-treatment baseline. The primary endpoint is the brain metabolic effects of treatment with CNM-Au8 as assessed by an improvement of 31P-MRS assessment of Brain Tissue Cellular Redox Potential defined by the measured tissue ratio of NAD+:NADH concentrations following 12 weeks of once daily treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give written informed consent.
2. Male or female patients aged 35 years or greater (inclusive) and less than 75 years of age at the time of ALS diagnosis.
3. Patients with a confirmed ALS diagnosis: "definite ALS" or "probable ALS" or "possible" diagnostic criteria per the revised El Escorial Criteria as determined by a neurologist subspecializing in ALS (e.g., the Principal Investigator by study site).
4. Stable background therapy (e.g., stable dosing of riluzole within the prior 6-weeks) per Investigator discretion.
5. At the time of Screening disease duration less than or equal to 24-months from symptom onset OR within 12-moths of a confirmed ALS diagnosis.
6. Forced vital capacity (FVC) >/= 60% of predicted value as adjusted for gender, height, and age at the Screening Visit.
7. Patients who are ambulatory (e.g., normal ambulation, early ambulation difficulties, or walks with assistance) on the ALSFRS-R scale.

Exclusion Criteria:

1. At Screening patients who utilize, or in the Investigator's judgment will be imminently dependent upon during the course of this study:

   1. Non-invasive ventilation
   2. Gastrostomy (e.g., use of percutaneous endoscopic gastrostomy tube)
   3. Use of wheel chair
2. Patient who have previously undergone tracheostomy.
3. Patient with a history of significant other major medical condition based on the Investigator's judgment.
4. Based on the investigator's judgment, patients who may have difficulty complying with the protocol and/or study procedures.
5. Patient with clinically significant abnormalities in hematology, blood chemistry, ECG, or physical examination not resolved by the Baseline visit which according to Investigator can interfere with study participation.
6. Patient participating in any other investigational drug trial or using investigational drug (within 12 weeks prior to screening and thereafter)
7. Females who are pregnant or nursing or who plan to get pregnant during the course of this clinical trial or within 6 months of the end of this trial.
8. Positive screen for drugs of abuse or known alcohol abuse.
9. Women of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control during the study or for 6 months following completion of study participation.
10. Women with a positive pregnancy test, are lactating, or are planning to become pregnant during the study.
11. Patients with implanted metal objects in their body that may be affected by an MRI procedure.
12. Patients who are claustrophobic or otherwise unlikely to be able to complete the MRI scanning procedures.
13. Patients with a history of gold allergy.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in 31P-MRS Redox Ratio (NAD+/NADH) | At 12 Weeks
  Mean change in average NAD+/NADH measured brain Redox Ratio by treatment group

OTHER OUTCOMES:
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of NAD+ | At 12 Weeks
  Mean change in average CNS concentration of NAD+ [mmol/kg] by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of NADH | At 12 Weeks
  Mean change in average CNS concentration of NADH [mmol/kg] by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of ATP | At 12 Weeks
  Mean change in average CNS concentration of ATP [mmol/kg] (as internal reference) by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Phosphocreatine (PCr) | At 12 Weeks
  Mean change in average CNS concentration of PCr [mmol/kg] by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Intracellular Inorganic Phosphate (Pi(in)) | At 12 Weeks
  Mean change in average CNS concentration of Pi(in) [mmol/kg] by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Extracellular Inorganic Phosphate (Pi(ex)) | At 12 Weeks
  Mean change in average CNS concentration of Pi(ex) [mmol/kg] by treatment group
Mean Change in 31P-MRS Bioenergetic Metabolite CNS Tissue Concentration of Uridine Diphosphate Glucose (UDPG) | At 12 Weeks
  Mean change in average CNS concentration of UDPG [mmol/kg] by treatment group
Mean Change in 31P-MRS Membrane Component Tissue Concentration of Phosphoethanolamine (PE) | At 12 Weeks
  Mean change in average CNS concentration of PE [mmol/kg] by treatment group
Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Phosphocholine (PC) | At 12 Weeks
  Mean change in average CNS concentration of PC [mmol/kg] by treatment group
Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Glycerophosphoethanolamine (GPE) | At 12 Weeks
  Mean change in average CNS concentration of GPE [mmol/kg] by treatment group
Mean Change in 31P-MRS Membrane Component CNS Tissue Concentration of Glycerophosphocholine (GPC) | At 12 Weeks
  Mean change in average CNS concentration of GPC [mmol/kg] by treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Elliott, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No